CLINICAL TRIAL: NCT06429098
Title: Study of A Venetoclax-based, Anthracycline-free Regimen in Patients With Newly Diagnosed CBFβ::MYH11-positive Acute Myeloid Leukemia
Brief Title: Study of A Venetoclax-based, Anthracycline-free Regimen in Newly Diagnosed CBFβ::MYH11(+) AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023371
Record Dates: First submitted 2024-05-14; First posted 2024-05-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: venetoclax; acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine; Decitabine; Cytarabine; 1-beta-D-arabinofuranosylcytosine 5'-monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax, Azacitidine/Decitabine/, Cytarabine (Experimental): INDUCTION: Patients receive 2 cycles of VEN/HMA as induction therapy. Venetoclax orally (PO) once daily (QD) on days 1-28, azacitidine subcutaneously (SC) on days 1-7 or decitabine intravenously (IV) over 30-60 minutes on days 1-5.
  CONSOLIDATION: Fit patients will receive four cycles of consolidation therapy with high-dose cytarabine (2g/m2 every 12 hours, on days 1-3) combined with venetoclax (on days 1-7). Unfit patients will continue to receive VEN/HMA until disease progression.
  Interventions: Drug: Venetoclax; Drug: azacitidine; Drug: decitabine; Drug: Cytarabine

INTERVENTIONS:
Drug: Venetoclax — Given PO, once daily. Treatment in cycle 1, the dose is 100 mg on day 1, then ramp up to 400mg. In all subsequent cycles, the dose of venetoclax is initiated at 400 mg daily.
  Other Names: ABT-199; ABT199; Venclexta
Drug: azacitidine — Given SC
  Other Names: 5 AZC; 5-AZC
Drug: decitabine — Given IV
  Other Names: Dacogen
Drug: Cytarabine — Given IV
  Other Names: 1-.beta.-Cytosine arabinoside; Ara-C

SUMMARY:
This investigator-initiated, single-arm, phase II trial is aimed to evaluate the efficacy and safety of a venetoclax-based, anthracycline-free regimen in patients with newly diagnosed CBFβ::MYH11-positive acute myeloid leukemia.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the CR (complete remission) / CRi (complete remission with incomplete blood count recovery) rate of 2 cycles of VEN/HMA in patients with newly diagnosed (ND) CBFβ::MYH11-positive acute myeloid leukemia(AML).

Secondary Objectives:

1. To determine the overall response rate (ORR) of 2 cycles of VEN/HMA in patients with ND CBFβ::MYH11-positive AML.
2. To determine the safety of the combination regimen.
3. To study the trajectories of molecular measurable residual disease (MRD) during the therapy.
4. To evaluate the impact of baseline genomic alterations on response and survival of the combination regimen.
5. To assess the duration of response, overall survival (OS) and event free survival (EFS) of patients.

OUTLINE:

INDUCTION:

Patients with newly diagnosed CBFβ::MYH11(+) AML receive 2 cycles of VEN/HMA as induction therapy. Venetoclax orally (PO) once daily (QD) on days 1-28, azacitidine subcutaneously (SC) on days 1-7 or decitabine intravenously (IV) over 30-60 minutes on days 1-5.

CONSOLIDATION:

Patient fitness will be reassessed according to the Ferrara criteria if CR or CRi is achieved after 2 cycles of VEN/HMA. Fit patients will receive four cycles of consolidation therapy with high-dose cytarabine (2g/m2 every 12 hours, on days 1-3) combined with venetoclax (on days 1-7). Unfit patients will continue to receive VEN/HMA until disease progression.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years.
2. Newly diagnosed CBFβ::MYH11(+) AML.
3. Performance status 0-3 on the Eastern Cooperative Oncology Group (ECOG) Scale.
4. Subject must voluntarily sign and date an informed consent, prior to the initiation of any screening or study-specific procedures.

Ferrara's criteria are used to determine whether a patient is unfit, and a patient is deemed unfit if at least one of the following criteria is met:

1. Age>75 years.
2. There are serious underlying heart, lung, kidney, liver complications.
3. There are active infections that do not respond to anti-infective therapy.
4. There is cognitive impairment.
5. Other comorbidities that the doctor determines are not suitable for intensive chemotherapy.

Exclusion Criteria:

1. Subject has received treatment with a hypomethylating agent and/or other chemotherapeutic agents either conventional or experimental or targeted drug therapy for AML (except oral hydroxyurea and/or leukocytometry to reduce white blood cell count).
2. Pregnant or lactating women.
3. To the knowledge of the subject and investigator, subject may not be able to complete all study visits or procedures required by the study protocol, including follow-up visits, and/or be unable to comply with the required study procedures.
4. Other conditions deemed unsuitable for participation in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
composite complete remission rate | after 2 cycles of induction therapy with VEN/HMA (each cycle is 28 days).
  CR/CRi rate will be determined.

SECONDARY OUTCOMES:
Overall response rate (ORR) | after 2 cycles of induction therapy with VEN/HMA (each cycle is 28 days).
  ORR will be determined.
Incidence of adverse events | From the start of treatment until death or last follow-up, assessed for up to 3 years.
  Safety profile based on NCI CTCAE version 5.0 will be determined.
measurable residual disease (MRD) negativity | From the start of treatment until death or last follow-up, assessed for up to 3 years.
  MRD will be assessed by real-time qRCR.
Impact of concurrent gene mutations | Baseline
  The impact of concurrent gene mutations ( analysis via an 81-gene institutional next-generation sequencing platform) on response and the survival of the combination regimen will be assessed.
Overall survival (OS) | From the start of treatment until death or last follow-up, assessed for up to 3 years.
  OS will be assessed.
Event-free survival (EFS) | up to 3 years.
  EFS will be assessed.
Duration of response (DOR) | up to 3 years.
  DOR will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (2):
- China (2):
  - Ethical Committee of the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No